CLINICAL TRIAL: NCT04058236
Title: Glycocalyx Levels in Patients Undergoing Pancreatectomy With Human Albumin 5% vs. Gelofusine
Brief Title: Glycocalyx Levels in Patients Undergoing Pancreatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Consultant Anaesthesiologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1237-9121
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Endothelial Degeneration; Pancreatic Cancer; Pancreatectomy; Postoperative Pancreatic Fistula
Keywords: Glycocalyx levels; pancreatectomy; human albumin 5%; gelofusine; pancreatic fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula | interventions — Polygeline

STUDY DESIGN:
Intervention Model Description: Randomized control trial with Albumin 5% given as the intervention and Gelofusine as active control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized concealed assignment into 2 groups in opaque envelopes will be opened by care provider. Anaesthetic and ICU notes must not be revealed to outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human albumin 5% (Experimental): 10 patients with pancreatic cancer will receive human albumin 5% in a restrictive goal directed fluid regime preoperatively for the first 24 hours.
  Interventions: Other: human albumin 5%
- gelofusine (Active Comparator): 10 patients with pancreatic cancer will receive gelofusine in a restrictive goal directed fluid regime preoperatively for the first 24 hours.
  Interventions: Other: gelofusine.

INTERVENTIONS:
Other: human albumin 5% — Human Albumin 5% will be given as fluid management for this group in accordance to goal directed therapy and guided by stroke volume variation of approximately 12-15%. This percentage of SVV has been validated as a threshold above which fluid administration increases stroke volume with an area under the receiver operating characteristics curve reported at 0.87. If the SVV remains more than 15% for more than 2 minutes, 250ml of fluid replacement according to patient group will be given. These boluses are given in aliquots over 30 min to avoid effects of rapid volume expansion. and the same fluid and technique will be carried out within 24 hours intra and post operatively in the Intensive Care Unit (ICU). All clinical parameters and fluids including blood that will be given will be recorded.
  Other Names: Fluid management
  Arms: human albumin 5%
Other: gelofusine. — Gelofusine will be given as fluid management for this group in accordance to goal directed therapy and guided by stroke volume variation of approximately 12-15%. This percentage of SVV has been validated as a threshold above which fluid administration increases stroke volume with an area under the receiver operating characteristics curve reported at 0.87. If the SVV remains more than 15% for more than 2 minutes, 250ml of fluid replacement according to patient group will be given. These boluses are given in aliquots over 30 min to avoid effects of rapid volume expansion. and the same fluid and technique will be carried out within 24 hours intra and post operatively in the Intensive Care Unit (ICU). All clinical parameters and fluids including blood that will be given will be recorded.
  Other Names: Fluid management
  Arms: gelofusine

SUMMARY:
Background:

On the surface of every healthy cellular membrane resides a layer known as the glycocalyx. This structure consists of extracellular domains of receptor, adhesion and transmembrane molecules such as syndecan-1 covalently bound to highly negatively charged glycosaminoglycans, heparan sulfates. It has a principal role to maintain wall integrity, avoid inflammation and tissue oedema in vessels but in contrast, glycocalyx is robust and elevated on cancer cells. This study examines whether the endothelial glycocalyx layer is preserved in patients undergoing pancreatectomy with human albumin 5% vs. gelofusine in a restrictive goal directed fluid regime perioperatively for the first 24hours. Degradation of glycocalyx will be investigated by analyzing basic levels of the core protein syndecan-1 and heparan sulfates with post-operative samples.

DETAILED DESCRIPTION:
This is a prospective study that will be conducted in the Main Operating theatres of UMMC on patients with pancreatic cancer undergoing elective pancreatectomy (includes all forms of pancreatectomy such as Whipple's procedure, total or distal pancreatectomy).

This study aim to determine the association of glycocalyx degradation by measuring levels of syndecan-1 and heparan sulfate with type of colloidal fluid given, human albumin 5% versus gelofusine in a restrictive goal directed fluid therapy in pancreatectomy.

Institutional ethics approval and registration in Clinical Trial Registry will be obtained before recruiting the first case.

Recruited patients will be randomly allocated to either the group receiving human albumin 5% or gelofusine.

Sample size:

There is no previously published literature related exactly to the pathology and methods of this proposed study. Therefore, a preliminary sample size calculation will be based on the closest study on fluids with a two-sided confidence interval of 0.95 and a desired power of 0.80 to yield a result that investigators need nine patients in each group. After adjusting for drop out rate of 10%, investigators will recruit ten in each group for human albumin 5% and gelofusine respectively within the study period of 2 years.

Data collection:

1. Intraoperative phase All preoperative preparation including fasting will be done in accordance to UMMC protocol. Intraoperative monitoring includes standard routine monitoring as per American Society of Anaesthesiologist Guidelines, invasive haemodynamic monitoring with arterial blood pressure incorporating FloTrac, BIS and neuromuscular monitoring. All patients will be under general anesthesia.

   Fluid management for both groups are in accordance to goal directed therapy and guided by stroke volume variation of approximately 12-15%. If SVV is > 15%, 250ml of fluid replacement according to patient group will be given over 30 min within 24 hours intra and post operatively in the Intensive Care Unit (ICU). In both groups, all clinical parameters and fluids including blood that will be given will be recorded.
2. Post-operative phase:

   The allocated colloid fluid will be continued.

   Patients will be assessed for pancreatic fistula leak. The grading of pancreatic fistula will be defined according to the guideline of Revised 2016 International Study Group on Pancreatic Fistula (ISGPF).

   Reviews will be done on post op days 1, 3, 5 and 30. Amylase levels from drain tube post-op Day 3, 5 and 7 will be measured. The total duration of stay in intensive care, hospital and rate of mortality/ morbidity (re-laparotomy/ re-admission to ICU/ sepsis) within 30 days after surgery will be assessed and recorded.
3. Laboratory phase Blood samples are collected at 5 time points, a) preoperative, b) immediate postoperative and c) 24 hours postoperative d) Day 3 and e) Day 7 postoperative from both groups. The serum fraction will be frozen and stored at -80°C until assayed. Syndecan 1 concentrations and heparan sulfate concentrations are quantified using special enzyme-linked immunosorbent assay kit as previously reported. Inflammatory markers Interleukin-1 and CRP and any blood investigations as per hospital sepsis protocol will be determined as well.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* patients aged between 18-75 years old with written informed consent

Exclusion Criteria:

* Patients who refuse to participate,
* Have severe congestive heart failure (NYHA class III/IV) or severe respiratory disease (PaO2/FiO2 < 200),
* Suffer significant renal or hepatic dysfunction (creatinine raised >50 % or liver enzymes >50 % of normal values),
* Pregnant
* Allergic to gelofusine and human albumin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurence of pancreatic fistula leak | Within post-op 30 days
  Review will be done according to guideline of Revised 2016 International Study Group on Pancreatic Fistula (ISGPF)
Changes in serum syndecan 1 concentrations | Within post-op 7 days
  Blood samples are collected to check for syndecan 1 concentrations in serum
Changes in serum heparan sulfate concentrations | Within post-op 7 days
  Blood samples are collected to check for heparan sulfate concentrations in serum

SECONDARY OUTCOMES:
Changes in levels of Inflammatory markers Interleukin-1 and CRP | Within post-op 7 days
  Blood samples are collected to check level of the Inflammatory markers Interleukin-1 and CRP

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, MBBS, MMed, Principal Investigator — University Malaya, Malaysia
Locations (1):
- Anaesthesia Department, Faculty of Medicine, University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pries AR, Kuebler WM. Normal endothelium. Handb Exp Pharmacol. 2006;(176 Pt 1):1-40. doi: 10.1007/3-540-32967-6_1. PMID 16999215
- [Background] Woodcock TE, Woodcock TM. Revised Starling equation and the glycocalyx model of transvascular fluid exchange: an improved paradigm for prescribing intravenous fluid therapy. Br J Anaesth. 2012 Mar;108(3):384-94. doi: 10.1093/bja/aer515. Epub 2012 Jan 29. PMID 22290457
- [Background] Curry FE, Adamson RH. Endothelial glycocalyx: permeability barrier and mechanosensor. Ann Biomed Eng. 2012 Apr;40(4):828-39. doi: 10.1007/s10439-011-0429-8. Epub 2011 Oct 19. PMID 22009311
- [Background] Tarbell JM, Cancel LM. The glycocalyx and its significance in human medicine. J Intern Med. 2016 Jul;280(1):97-113. doi: 10.1111/joim.12465. Epub 2016 Jan 8. PMID 26749537
- [Background] Lobo DN, Bostock KA, Neal KR, Perkins AC, Rowlands BJ, Allison SP. Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet. 2002 May 25;359(9320):1812-8. doi: 10.1016/S0140-6736(02)08711-1. PMID 12044376
- [Background] Chappell D, Bruegger D, Potzel J, Jacob M, Brettner F, Vogeser M, Conzen P, Becker BF, Rehm M. Hypervolemia increases release of atrial natriuretic peptide and shedding of the endothelial glycocalyx. Crit Care. 2014 Oct 13;18(5):538. doi: 10.1186/s13054-014-0538-5. PMID 25497357
- [Background] Sulzer JK, Sastry AV, Meyer LM, Cochran A, Buhrman WC, Baker EH, Martinie JB, Iannitti DA, Vrochides D. The impact of intraoperative goal-directed fluid therapy on complications after pancreaticoduodenectomy. Ann Med Surg (Lond). 2018 Oct 16;36:23-28. doi: 10.1016/j.amsu.2018.10.018. eCollection 2018 Dec. PMID 30370053
- [Background] Jacob M, Bruegger D, Rehm M, Stoeckelhuber M, Welsch U, Conzen P, Becker BF. The endothelial glycocalyx affords compatibility of Starling's principle and high cardiac interstitial albumin levels. Cardiovasc Res. 2007 Feb 1;73(3):575-86. doi: 10.1016/j.cardiores.2006.11.021. Epub 2006 Nov 21. PMID 17196565
- [Background] Alphonsus CS, Rodseth RN. The endothelial glycocalyx: a review of the vascular barrier. Anaesthesia. 2014 Jul;69(7):777-84. doi: 10.1111/anae.12661. Epub 2014 Apr 28. PMID 24773303
- [Background] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Background] Myburgh JA, Finfer S, Bellomo R, Billot L, Cass A, Gattas D, Glass P, Lipman J, Liu B, McArthur C, McGuinness S, Rajbhandari D, Taylor CB, Webb SA; CHEST Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Hydroxyethyl starch or saline for fluid resuscitation in intensive care. N Engl J Med. 2012 Nov 15;367(20):1901-11. doi: 10.1056/NEJMoa1209759. Epub 2012 Oct 17. PMID 23075127
- [Background] Vincent JL, Russell JA, Jacob M, Martin G, Guidet B, Wernerman J, Ferrer R, McCluskey SA, Gattinoni L. Albumin administration in the acutely ill: what is new and where next? Crit Care. 2014 Jul 16;18(4):231. doi: 10.1186/cc13991. PMID 25042164
- [Background] Cooper DJ, Myburgh J, Heritier S, Finfer S, Bellomo R, Billot L, Murray L, Vallance S; SAFE-TBI Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Albumin resuscitation for traumatic brain injury: is intracranial hypertension the cause of increased mortality? J Neurotrauma. 2013 Apr 1;30(7):512-8. doi: 10.1089/neu.2012.2573. Epub 2013 Mar 21. PMID 23194432
- [Background] Finfer S, Bellomo R, Boyce N, French J, Myburgh J, Norton R; SAFE Study Investigators. A comparison of albumin and saline for fluid resuscitation in the intensive care unit. N Engl J Med. 2004 May 27;350(22):2247-56. doi: 10.1056/NEJMoa040232. PMID 15163774
- [Background] Kang H, Wu Q, Sun A, Liu X, Fan Y, Deng X. Cancer Cell Glycocalyx and Its Significance in Cancer Progression. Int J Mol Sci. 2018 Aug 22;19(9):2484. doi: 10.3390/ijms19092484. PMID 30135409